CLINICAL TRIAL: NCT05186012
Title: A Phase Ib/II Study of APG-1252 as a Single Agent or in Combination With Other Therapeutic Agent in Patients With Relapsed and/or Refractory Non-Hodgkin Lymphoma(NHL)
Brief Title: APG-1252 Monotherapy or in Combination With Other Therapeutic Agent in Subjects With Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APG1252LC101
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-08

CONDITIONS: NHL, Adult
Keywords: APG-1252
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — pelcitoclax; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Single agent) (Experimental)
  Interventions: Drug: APG-1252
- Arm B (combo) (Experimental)
  Interventions: Drug: APG-1252; Drug: Chidamide

INTERVENTIONS:
Drug: APG-1252 — APG-1252 administered via intravenous infusion for 30 minutes weekly (Day 1, 8, 15, 22).Every 28 days as a cycle.
  Other Names: Pelcitoclax
Drug: Chidamide — Chidamide 30mg orally BIW. Every 28 days as a cycle.
  Arms: Arm B (combo)

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetic, pharmacodynamic and efficacy of APG-1252 single agent and in combination with other therapeutic agent in patients with NHL.

DETAILED DESCRIPTION:
This is an open-label, multi-center Phase Ib/II study of safety, PK, PD and efficacy of APG-1252 as a single agent in relapsed/refractory NHL or in combination with chidamide in relapsed/refractory peripheral T cell lymphomas (PTCL) patients. The primary objective is to evaluate the safety and tolerability, identify dose-limiting toxicities (DLT), the maximum tolerated dose (MTD) and the recommended dose (RP2D) of APG-1252 monotherapy or in combination with chidamide in relapsed/refractory PTCL patients.

This study consists of two parts: The first part is the APG-1252 single agent cohort, including dose escalation phase with a standard 3+3 design and dose expansion phase with 6-15 patients at MTD dose level. The second part is the APG-1252 plus chidamide, including dose escalation phase with a standard 3+3 design and dose expansion phase with 9-12 patients at MTD dose level.

Patients will be treated in 28-day cycles. APG-1252 will be administered via intravenous infusion for 30 minutes weekly (Day 1, 8, 15, 22). Chidamide will be administered 30mg orally BIW. All subjects will continue to receive treatment until disease progression, unacceptable toxicities, or other treatment discontinuation criteria defined by the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Life expectancy ≥ 3 months.
2. Eastern Cooperative Oncology Group (ECOG) 0-1.
3. Corrected QT interval (QTcB or QTcF ) ≤ 450ms (male), or ≤ 470ms (female).
4. Patients with relapsed/refractory NHL in Part 1 (excluding Burkitt's lymphoma, lymphoblastic lymphoma, chronic lymphocytic leukemia/small lymphocytic lymphoma or primary central nervous system lymphoma) and relapsed/refractory PTCL in Part 2, previously treated with at least 1 prior line of therapy.
5. Patients must have an adequate bone marrow function.
6. Adequate hepatic, renal and coagulation function.
7. Male and female subjects of childbearing potential who agree to use highly effective methods of birth control during the period of therapy and for 90 days after the last dose of study drug.
8. Ability to understand and voluntarily sign a written informed consent form before performing any study procedures.
9. Compliance to study procedures.

Exclusion Criteria:

1. Prior history of allogeneic cell transplant, adoptive cellular immunotherapy within 2 years, or autologous hematopoietic stem cell transplantation within 6 months prior to the first dose.
2. Monoclonal antibody therapy within 4 weeks prior to the first dose.
3. Received anti-cancer therapy within 14 days prior to the first dose of therapy, including chemotherapy, radiotherapy, immunotherapy or hormone therapy for anti-tumor purposes; or 28 days for any investigational agent prior to the first dose of therapy.
4. Continuance of toxicities due to prior radiotherapy or chemotherapy agents that do not recover to ≤ Grade 1 except alopecia or neuropathy.
5. Not recovered from recent surgical procedures based on investigator's discretion. Major surgical procedure within ≤28 days or minor surgical procedure (excluding biopsy) within ≤14 days prior to initiating study treatment.
6. Prior exposure to BCL-xL inhibitor. Subjects who have been treated with chidamide can still be included in the study unless they were intolerant.
7. Intolerant to other Bcl-2 family protein inhibitors.
8. Has known central nervous system (CNS) involvement or the prior history of primary central nervous system lymphoma.
9. Prior history of cardiovascular disease ≥ grade 2 (New York Heart Association grade 2 cardiovascular disease is defined as that the patient feels comfortable at rest, but ordinary physical activities lead to fatigue, palpitation, dyspnea or angina pectoris). Unstable angina, myocardial infarction, or coronary revascularization within 180 days prior to the first dose.
10. Use of therapeutic doses of anti-coagulants is an exclusion, including anti-platelet agents. Use of low-dose anticoagulation medications to maintain the patency of a central intravenous catheter is permitted. Aspirin taken within 1 week before the first dose is an exclusion.
11. Known bleeding diathesis/disorder. Recent history of non-chemotherapy induced thrombocytopenia associated a major bleeding episode or a history of being refractory to platelet transfusions within 1 year prior to the first dose. Gastrointestinal bleeding or active peptic ulceration within 3 months prior to the first dose. Active immune thrombocytopenic purpura (ITP), active autoimmune hemolytic anemia (AIHA).
12. A potentially bleeding condition or the presence of clinically significant bleeding signs.
13. Known to be allergic to the drug component or its analogues.
14. Pregnancy or lactation, or pregnancy is expected during the study period or within 3 months after the last administration of treatment.
15. Within 3 years before entering the study, the subject had a history of active malignant tumors other than NHL, except that: Fully treated cervical carcinoma in situ; Completely resected basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; Confinement and resection of previously cured malignancies (or other treatment).
16. Uncontrolled systemic infections (viruses, bacteria, or fungi), including but not limited to Covid-19 RNA positive, HBV-SURFACE antigen positive and HBV-DNA≥2,000 copies/mL or ≥500 IU/ mL; Hepatitis C virus (HCV) antibody positive; human immunodeficiency virus (HIV) antibody positive.
17. A significant history of renal, neurological, psychiatric, pulmonary, endocrine, metabolic, immune, cardiovascular or liver disease. The investigator believes that participating in this study will have an adverse effect on him / her.
18. Uncontrolled other clinically significant symptoms, including but not limited to uncontrolled serious infection, febrile neutropenia occured within 1 week before administration. Symptomatic congestive heart failure, unstable angina, arrhythmia, or social environment that may affect study compliance.
19. Any other condition or circumstance that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 28 days
  DLT will be defined based on the rate of drug-related grade 3-5 adverse events experienced within the first 28 days of study treatment. These will be assessed via CTCAE version 5.0.
Maximally tolerated dose (MTD) | 28 days
  MTD will be determined based on DLTs observed during the first 28 days of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Chair — Ascentage Pharma Group Inc.
Locations (4):
- China (4):
  - Henan Provincial Oncology Hospital, Zhengzhou, Henanan
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Jiangsu Province Hospital, Nanyang
  - Shanghai Jiao Tong University school of medicine Ruijin Hospital, Shanghai